CLINICAL TRIAL: NCT03785496
Title: Phase II Study to Evaluate Efficacy of PDR001 in Patients With Squamous Cell Carcinoma of the Esophagus
Brief Title: Study to Evaluate Efficacy of PDR001 in Patients With Squamous Cell Carcinoma of the Esophagus
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2018-0938
Record Dates: First submitted 2018-12-06; First posted 2018-12-24 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Histologically Confirmed Unresectable or Metastatic Squamous Cell Carcinoma of the Esophagus Who Failed on Standard Treatment
MeSH Terms: interventions — spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PDR001 (Experimental): PDR001 will be administered once every 3 weeks via i.v. infusions over 30 minutes, respectively. Infusions of each antibody can be extended to up to 2 hours if clinically indicated. A scheduled dose of ongoing study drugs may be delayed by up to 7 days to recover from previous AEs or a missed visit. If a scheduled dose of ongoing study drugs is delayed longer than 7 days due to an unresolved AE, the administration should be skipped and treatment resumed at the next scheduled dose. The assessment schedule will be shifted accordingly.
  Interventions: Drug: PDR001

INTERVENTIONS:
Drug: PDR001 — PDR001 will be administered once every 3 weeks via i.v. infusions over 30 minutes, respectively. Infusions of each antibody can be extended to up to 2 hours if clinically indicated. A scheduled dose of ongoing study drugs may be delayed by up to 7 days to recover from previous AEs or a missed visit. If a scheduled dose of ongoing study drugs is delayed longer than 7 days due to an unresolved AE, the administration should be skipped and treatment resumed at the next scheduled dose. The assessment schedule will be shifted accordingly.

SUMMARY:
Single arm phase II PDR001( 300mg, IV) will be treated every 3 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed squamous cell carcinoma of the esophagus
2. Age ≥ 20
3. ECOG PS 0-2
4. Ineligibility for local therapy (surgery or radiotherapy), including but not limited to:

   * Patients with distant metastases (stage M1, stage IVB)
   * Patients with disease progression and/or recurrence after chemoradiotherapy
   * Patients with disease recurrence after surgical excision for primary esophageal cancer
   * Ineligible patient for surgery and/or CCRT due to medical condition
   * Ineligible patients with T4b for surgery and/or CCRT due to invasive organs such as large vessels, heart
5. Prior palliative chemotherapy including platinum-based chemotherapy. When recurred within 6 months of definitive/neoadjuvant/adjuvant chemo-, the chemotherapy is considered a line of therapy
6. At least one uni-dimensionally measurable disease as defined by RECIST ver 1.1
7. Adequate organ function for treatment (Table 1)
8. 12-Lead electrocardiogram (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
9. QTcF interval ≤470 msec and without history of Torsades de Pointes or other symptomatic QTcF abnormality
10. LVEF (by MUGA or echocardiogram) of ≥50%
11. The patient has provided signed informed consent
12. System Laboratory Value :Hematological

    * Absolute neutrophil count (ANC) ≥1,500 /mcL
    * Platelets ≥100,000 / mcL Hemoglobin ≥9 g/dL or ≥5.6 mmol/L without transfusion orErythropoietin(EPO) dependency (within 7 days of assessment).
    * Renal Serum creatinine OR Measured or calculated creatinine clearance(GFR can also be used in place of creatinine or CrCl) ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN
    * Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN
    * Aspartate transaminase(AST)(SGOT) and Alanine Aminotransferase(ALT)(SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases -Albumin >2.5 mg/dL
    * Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT)
    * Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants a Creatinine clearance should be calculated per institutional standard.

Exclusion Criteria:

1. Presence of symptomatic CNS metastases, or CNS metastases that require local CNS-directed therapy (such as radiotherapy or surgery). Patients with treated brain metastases should be neurologically stable (for 4 weeks post treatment and prior to study enrollment) and off of steroids for at least 2 weeks before administration of any study drug.
2. Previous treatment with anti- PD-1, and/or PD-L1
3. Two or more previous systemic cytotoxic chemotherapy (chemotherapy administered with concurrent radiotherapy for local control is not counted)
4. Any major operation within 4 weeks of baseline disease assessment
5. Any medical condition that would, in the investigator's judgement, prevent the patient's participation in the clinical study due to safety concerns, compliance with clinical study procedures or interpretation of study results, including but not limited to:

   * Prior immune-related adverse events requiring treatment discontinuation
   * Ongoing symptomatic interstitial lung disease (ILD), noninfectious pneumonitis or history of drug induced interstitial lung disease
6. Impaired cardiac function or clinically significant cardiac disease, including any of the following:

   * Clinically significant and/or uncontrolled heart disease such as congestive heart failure requiring treatment (NYHA Grade ≥ 2), uncontrolled hypertension or clinically significant arrhythmia
   * QTcF > 470 msec on screening ECG or congenital long QT syndrome
   * Acute myocardial infarction or unstable angina pectoris < 3 months prior to study entry
7. Active infection, including active tuberculosis requiring systemic antibiotic therapy
8. Known human immunodeficiency virus (HIV) infection (no testing required).
9. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection, or HBV/HCV carriers/infections requiring antiviral treatment (testing required)
10. Use of any live vaccines against infectious diseases (e.g. varicella, pneumococcus) within 4 weeks of initiation of study treatment.
11. Major surgery within 2 weeks of the first dose of study treatment (mediastinoscopy, insertion of a central venous access device, and insertion of a feeding tube are not considered major surgery).
12. Radiotherapy within 4 weeks of the first dose of study drug except palliative radiation to painful bony lesion (this must comprise less than 30% of the bone marrow) at least 2 weeks prior to the first dose of study drug.
13. Systemic anti-cancer therapy within 2 weeks or 5 x T ½, whichever is longer of the first dose of study treatment. For cytotoxic agents that have major delayed toxicity, e.g. mitomycin C and nitrosoureas, 4 weeks is indicated as washout period. For patients receiving CTLA-4 antagonists, 6 weeks is indicated as the washout period
14. Presence of ≥ CTCAE Grade 2 toxicity (except alopecia, peripheral neuropathy and ototoxicity, which are excluded if ≥ CTCAE Grade 3) due to prior cancer therapy
15. Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumors treated curatively and without evidence of recurrence for at least 5 years prior to study entry.
16. Pregnant or lactating women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
17. Patients receiving concomitant immunosuppressive agents or chronic corticosteroids (≥10 mg of prednisone or equivalent) at the time of first study dose
18. Other severe acute or chronic medical condition or laboratory abnormality that may increase the risk associated with trial participation
19. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 150 days after the last dose of PDR001. Highly effective contraception methods include:

    * Total abstinence (when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) total hysterectomy or tubal ligation at least 1.5 months before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female patients on the study the vasectomized male partner should be the sole partner for that patient.
    * Use of oral, injected or implanted hormonal methods of contraception or placement of an intrauterine device (IUD) or intrauterine system (IUS), or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.

    In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment. Women are considered post-menopausal and not of child bearing potential if they have had over 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile age appropriate (e.g. generally 40-59 years), history of vasomotor symptoms (e.g. hot flushes) in the absence of other medical justification or have had surgical bilateral oophorectomy (with or without hysterectomy), total hysterectomy, or tubal ligation at least 1.5 months ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow-up hormone level assessment is she considered not of child bearing potential.
20. Sexually active males unless they use a condom during intercourse while taking treatment and for 150 days after the last dose of PDR001. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate efficacy of PDR001 by Objective Response rate by RECIST(Response Evaluation Criteria In Solid Tumors) | Repeated tumor imaging will be performed every 2 cycle (each cycle is 21 days) after baseline imaging
  In the first stage of the trial, 22 patients will be recruited, and their tumor response will be assessed RECIST criteria, which is widely used tumor assessment criteria in immuno-oncology agent trials. The best response until 6 months according to irRECIST will be evaluated, and this trial will proceed to second stage if three or more respondents (irPR or irCR) are observed among 22 patients. The response (PR or CR) should be confirmed by next disease assessment(6 weeks/2cycles after initial response).
  Subjects who discontinue trial treatment for a reason other than recurrence will move into the Follow-Up Phase and should be assessed every 16 weeks (± 14 days) by radiologic imaging to monitor disease status.

SECONDARY OUTCOMES:
To evaluate antitumor efficacy of PDR001: PFS(Progression-Free Survival) | Biopsies will be taken during the screening period (e.g., within 7 days before treatment [pre-dose]), on treatment (Day 22 of first dose) and post-treatment (e.g., within 28 days after progression)
  PFS is defined as the time between the day of first cycle and the date of first documentation of progression or date of death, whichever occurs first. Documentation of progression will be defined as per RECIST criteria based on investigator assessment. Patients without documented progression or death will be censored at the date of last tumor assessment (or, if no tumor assessments are performed after the baseline visit).
To evaluate antitumor efficacy of PDR001: OS(Overall survival) | Biopsies will be taken during the screening period (e.g., within 7 days before treatment [pre-dose]), on treatment (Day 22 of first dose) and post-treatment (e.g., within 28 days after progression)
  OS is defined as the time between the day of first cycle and the date of death. Patients without documented death will be censored at the date of last contact.
To evaluate antitumor efficacy of PDR001 | Biopsies will be taken during the screening period (e.g., within 7 days before treatment [pre-dose]), on treatment (Day 22 of first dose) and post-treatment (e.g., within 28 days after progression)
  DCR is defined as the percentage of patients with cancer who have achieved complete response, partial response and stable disease to a therapeutic intervention in clinical trials of anticancer agents. RECIST will be used in this study for assessment of tumor response. While either CT or MRI may be utilized, as per RECIST, CT is the preferred imaging technique in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Byoung Chul Cho, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee DK, Park SR, Kim YH, Lee YG, Shin SJ, Ahn BC, Lee SS, Lim SM, Kim HR, Cho BC, Hong MH. A phase 2 study of spartalizumab (PDR001) among patients with recurrent or metastatic esophageal squamous cell carcinoma (KCSG HN18-17, K-MASTER project 12). Oncoimmunology. 2024 Jun 24;13(1):2371563. doi: 10.1080/2162402X.2024.2371563. eCollection 2024. PMID 38919826